CLINICAL TRIAL: NCT00226590
Title: Phase II Trial of Induction Gemcitabine and Carboplatin Followed by Paclitaxel and Carboplatin With Concurrent Thoracic Radiation for Patients With Unresectable Stage IIIA/IIIB Non-Small Cell Lung Cancer
Brief Title: Induction Gemcitabine & Carboplatin Followed by Paclitaxel & Carboplatin +XRT in NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13240; 13189 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Results first posted 2011-05-23 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2011-05

CONDITIONS: Lung Cancer
Keywords: non-small cell lung cancer; carcinoma; unresectable; Stage IIIA; Stage IIIB; thoracic radiation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Gemcitabine; Carboplatin; Paclitaxel; Radiation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined Therapy (Experimental): In this trial we adopted the approach of using both induction and concurrent chemotherapy together with TRT planned conformally to a tumor dose of 74 Gy.
  Interventions: Drug: Gemcitabine; Drug: Carboplatin; Drug: Paclitaxel; Procedure: Radiation

INTERVENTIONS:
Drug: Gemcitabine — Induction Chemotherapy.
  Other Names: Gemzar
Drug: Carboplatin — Induction Chemotherapy. Weekly Carboplatin and Paclitaxel During Thoracic Radiation Therapy.
  Other Names: Paraplatin
Drug: Paclitaxel — Weekly Carboplatin and Paclitaxel During Thoracic Radiation Therapy.
  Other Names: Taxol
Procedure: Radiation — Radiation Therapy will begin on day 57 if there has been adequate hematologic recovery from Induction Chemotherapy.
  Other Names: Radiation Therapy

SUMMARY:
This is a single institution Phase II study for patients with unresectable Stage IIIA and IIIB non-small cell lung cancer. The treatment started with 2 cycles of gemcitabine and carboplatin followed by concurrent chemotherapy with radiation. The chemoradiation included using paclitaxel and carboplatin with daily thoracic radiation to a total dose of 74 Gy. Response rate was determined following the chemotherapy with gemcitabine and carboplatin and evaluated again after the chemoradiation. Treatment toxicities were also assessed.

DETAILED DESCRIPTION:
In this trial we adopted the approach of using both induction and concurrent chemotherapy together with Thoracic Radiation Therapy (TRT) planned conformally to a tumor dose of 74 Gy. Substitution of gemcitabine for paclitaxel in the induction chemotherapy allowed us to evaluate the impact of RRM1 expression on the activity of this agent. The expression of Ribonucleotide Reductase, M1 Subunit (RRM1) was evaluated prior to initiation of therapy, following induction chemotherapy but prior to concurrent chemoradiation, and following completion of all therapy by CT-guided core needle biopsies. This is a single institution phase II clinical trial, of induction treatment with gemcitabine and carboplatin followed by concurrent chemoradiation using paclitaxel and carboplatin and daily thoracic radiation to a total dose of 74 Gy for patients with unresectable Stage IIIA and IIIB NSCLC. The specific clinical objectives of this study are as follows: To determine the response rate (both CT scan and PET scan assessment) to two cycles of induction chemotherapy with gemcitabine and carboplatin; To determine the response rate (both CT scan and PET scan assessment) to concurrent thoracic radiation and weekly paclitaxel and carboplatin; To evaluate the patterns of local and distant failure for patients treated with induction chemotherapy followed by concurrent chemoradiation according to this regimen; To estimate the median, 1 year, and overall survival; To assess acute and long term toxicities of treatment.

ELIGIBILITY:
Eligibility Criteria:

* Histologically confirmed unresectable non-small cell carcinoma of the lung (adenocarcinoma, squamous cell carcinoma or anaplastic large cell carcinoma). See below for TNM eligibility. Mediastinoscopy or thoracoscopy in patients with mediastinal lymph node enlargement of < 2 cm on CT scans of suspicious on PET scan to confirm suspected involvement. These staging procedures are not mandatory for patients with obvious nodal involvement (2.0 cm or greater). Staging system: The New International Staging System for lung cancer (Clifton F. Mountain, 1997) will be followed. The following stages will be eligible:
* Patients with stage IIIa disease will be eligible if it is felt that they are not candidates for possible resection following neo-adjuvant therapy (unresectable T3N1 or T1-3 primary tumors with metastasis limited to single station ipsilateral mediastinal lymph nodes). Patients with stage IIIb disease without significant* pleural effusion will be eligible. This includes patients with metastases to contralateral mediastinal or supraclavicular nodes.
* Patients without significant pleural effusion will constitute those in whom 1) it is seen on CT scan only or 2) does not reaccumulate after one thoracentesis and is cytologically negative.
* No evidence of distant metastasis.
* Patients must have measurable disease by the Recist Evaluation Criteria in Solid Tumors (RECIST) criteria. Baseline measurements/evaluations must be obtained within 4 weeks prior to registration.
* Patients must not have small cell carcinoma as part of the histological specimen (World Health Organization [WHO] classification 22.40)
* Performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1 at time of registration.
* Patients with preexisting clinically significant peripheral neuropathy are ineligible.
* Weight loss of ≤ 5% in the preceding three months
* No prior systemic chemotherapy or thoracic radiotherapy.
* Patients must have adequate bone marrow reserve as determined by the following laboratory values: Obtained within 14 days prior to registration.
* White blood cell count 4000/ul or greater and granulocyte count of 1500/ul or greater
* Platelet count of 100,000/ul or greater
* Hemoglobin of 10 gms/dl or greater.
* Adequate renal and liver function as determined by the following laboratory values: Obtained within 14 days prior to registration.
* Serum creatinine < 1.5 mg/dl or creatinine clearance greater than 50 cc/min
* Bilirubin less than 1.5 mg/dl
* SGOT less than 1.5 times normal
* No history of a prior or concomitant malignancy in the past five years except for surgically cured basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* No concomitant life threatening or uncontrolled serious medical illness such as cardiac arrhythmia, end stage congestive heart failure, liver disease with significant hepatic insufficiency, organic brain syndrome.
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception.
* Age greater than or equal to 18 years
* Written, informed consent must be obtained prior to registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Bepler, MD, PhD, Principal Investigator — Karmanos Cancer Institute (formerly at H. Lee Moffitt Cancer Center & Research Institute)
Locations (1):
- H. Lee Moffitt Cancer Center & Research Insitute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination Therapy: In this trial we adopted the approach of using both induction and concurrent chemotherapy together with TRT planned conformally to a tumor dose of 74 Gy.
Period: Overall Study
Arm/Group | Combination Therapy
Started | 39
Completed | 39
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Response Allowed Them to Proceed to Chemoradiation
Description: Response Rates - Complete Response (CR) + Partial Response (PR): We determined the number of participants whose response (both CT and PET assessment) to two cycles of induction chemotherapy with gemcitabine and carboplatin allowed them to proceed to chemoradiation. Response was evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.
Time Frame: Ranging from 2 weeks up to 4 years, 9 months
Population: Per Protocol
Measure: Number; unit: participants
Groups:
- Induction Therapy: Tolerance of Induction Therapy prior to Chemoradiation
Arm/Group | Induction Therapy
Number analyzed (Participants) | 39
participants | 38

2. Secondary Outcome: Progression Free Survival
Description: To determine median Progression Free Survival rate. Progression-free survival (PFS) is defined as the interval between the date of the first chemotherapy administration and the date of objective progression or death. Progression was evaluated using the new international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee.
Time Frame: Ranging from 2 weeks up to 4 years, 9 months
Population: per protocol
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 38
months | 22.7 [2.9 to 69.9]

3. Secondary Outcome: Overall Survival
Description: To determine median Overall Survival rate
Time Frame: Ranging from 2 weeks up to 4 years, 9 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination Therapy
Number analyzed (Participants) | 38
months | 14.3 [4.1 to 74.4]

4. Secondary Outcome: Treatment Completion
Description: The number of participants who completed all treatment on schedule without dose reductions or delays.
Time Frame: Ranging from 2 weeks up to 4 years, 9 months
Population: per protocol
Measure: Number; unit: participants
Arm/Group | Combination Therapy
Number analyzed (Participants) | 38
participants | 19

ADVERSE EVENTS:
Time Frame: Ranging from 2 weeks up to 4 years, 9 months
Arm/Group | Combination Therapy
Serious Adverse Events (participants affected / at risk) | 8/39
Other Adverse Events (participants affected / at risk) | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Therapy (N=39)
Esophageal stricture requiring dilatation (Gastrointestinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hydropneumo (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No